CLINICAL TRIAL: NCT00911456
Title: Can 3D Ultrasound Be Used Reproducibly by Radiation Therapists in Partial Breast Image-Guided Radiation Therapy?
Brief Title: Can 3D Ultrasound Be Used Reproducibly by Radiation Therapists in Partial Breast Image-Guided Radiation Therapy
Acronym: IGRT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: British Columbia Cancer Agency (Other)
Responsible Party: Tanya Berrang, British Columbia Cancer Agency
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0001
Record Dates: First submitted 2009-05-29; First posted 2009-06-02 (Estimated); Last update posted 2012-02-17 (Estimated); Status verified 2009-10

CONDITIONS: Radiation Therapy for Primary Breast Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Image-Guided Radiation Therapy using 3D Ultrasound Guided-Therapy — Subjects will have 3 x 3DUS during radiation therapy
Procedure: Ultrasound Guided Imaging — Subjects will undergo a CT scan and an US of your breast for the planning of radiation therapy after a breast conserving operation.
  About 1 week after the start of radiation treatment subjects will have a second CT and US. During this visit subjects will have one CT and three US's. These US's will be performed by 3 different radiation therapists. Part of the current study is to compare the similarity of the 3 US pictures taken by different individuals.
Procedure: 3 DUS — 3 DUS

SUMMARY:
To determine if the Clarity 3DUS (3D Ultrasound) system can be used by multiple individuals to acquire 3DUS images and produce consistent TB (Tumor Bed) shifts for breast IGRT (Image-Guided Radiation Therapy).

DETAILED DESCRIPTION:
TB Contouring The CT1, CT2, and US1 tumor beds will be manually contoured on the RM workstation by one of the study radiation therapists. Contouring will be performed using previously defined contouring guidelines. Available automatic contouring tools, including the 'interpolate' contouring function, may be utilized and contouring times will be recorded.

IGRT Assessment The patient will be set up on the breast board in treatment position. The 'ultra path' component of the Clarity system, which displays the path of the previous US acquired at CT simulation, will be used to guide the acquisition of US2. Although performed in the simulator room, the Clarity system will be used in 'treatment mode' thus simulating Clarity as it is used for IGRT. The study RT will first acquire the US2 scan. All steps following the acquisition of US2 will be performed off-line on the RM workstation without the need for further simulator or patient time.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be 27 consenting women undergoing CT simulation for adjuvant breast radiotherapy at VIC ≤16 weeks after BCS.
* Women must have primary tumors <3cm, pathologically N0 disease, and negative surgical margins.
* Seroma clarity score <2

Exclusion Criteria:

* Patients will be excluded if they have had mastectomy or receive adjuvant chemotherapy that results in the CT simulation session occurring >16 weeks after the BCS date.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2009-10; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Will the Clarity of breast IGRT product have the potential to improve localization through its ability to compare 3DUS at the time of planning to 3DUS at the time of treatment. | Outcome will be measured three times during the 3DUS

CONTACTS AND LOCATIONS:
Overall Officials: Tanya Berrang, Principal Investigator — British Columbia Cancer Agency
Locations (1):
- BC Cancer Agency Vancouver Island BCCA, Victoria, British Columbia, Canada